CLINICAL TRIAL: NCT05906173
Title: Successful International Training of Non-Technical Medical Crisis Skills Using Remote, Augmented Reality Simulation
Brief Title: Augmented Reality (AR) Chile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Thomas Caruso, Clinical Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 70882
Record Dates: First submitted 2023-06-07; First posted 2023-06-15 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Educational Problems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mixed Reality Simulation (Experimental): Participants in the experimental arm will be introduced to workplace training modules through an Augmented Reality (AR) headset.
  Interventions: Other: Augmented Reality (AR)

INTERVENTIONS:
Other: Augmented Reality (AR) — AR headset - a device that the participants will wear over their head and eyes and will add holographic elements to a live view of workplace training scenario

SUMMARY:
This is an international, collaborative study evaluating the non-technical skills (NTS) of anesthesiology residents. The goal is to explore the capability of performing a remote, international AR simulation for the purpose of assessing NTS during a neonatal medical crisis. Simulation experts in the United States will facilitate the AR simulations with anesthesiology residents in Chile. The medical simulation itself is grounded in traditional best practices in accordance with the American Heart Association and Neonatal Resuscitation Program.

ELIGIBILITY:
Inclusion Criteria:

* age above 18

Exclusion Criteria:

* a history of severe motion sickness
* currently have nausea, a history of seizures
* wear corrective glasses (they are not compatible with the AR hardware).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-08-10 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Individual performance of non-technical skills assessed by Anaesthetist Non-Technical Skills (ANTS) | immediately after simulation
  The Anaesthetist Non-Technical Skills (ANTS) tool previously published by Fletcher et al. translated in French. The ANTS scoring system uses four categories assessing task management, teamworking, situation awareness and decision-making (1 to 4 points by categories). The minimum score is 4 and the maximum 16

SECONDARY OUTCOMES:
Individual performance of non-technical skills assessed by Behaviorally Anchored Rating Scale (BARS) | immediately after simulation
  The BARS scoring system uses four categories assessing situation awareness, decision-making, communication and teamwork. The score ranges from 1 and 9 (1 = poor and 9 = excellent)
System Usability Scale (SUS) Score | immediately after simulation
  The scale has 10 items. Scores ranges from 1-5 (1 = strongly disagree and 5 = strongly agree)
ISO Ergonomic scale | immediately after simulation
  The scale has 6 items. Scores ranges from 1-5 (1 = strongly disagree and 5 = strongly agree)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Caruso, MD,PhD, Principal Investigator — Stanford University
Locations (1):
- Lucile Parkard Children's Hospital, Stanford, California, United States